CLINICAL TRIAL: NCT05598970
Title: Family and Childhood Development: Kizazi Kijacho ('The Next Generation') - a Cluster Randomised Controlled Trial
Brief Title: Family and Childhood Development: The Next Generation ('Kizazi Kijacho')
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Collaborators: EDI Global (Unknown); Elizabeth Glaser Pediatric AIDS Foundation (EGPAF) (Unknown); D-Tree International (Unknown); Ifakara Health Institute (IHI) (Unknown); Yale University (Other); University of Chile (Other); NHH-Norwegian School of Economics (Unknown); Chr. Michelsen Institute (Unknown)
Responsible Party: Principal Investigator, Ingvild Almås, Professor, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2022-01356-01
Record Dates: First submitted 2022-10-20; First posted 2022-10-31 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Parenting; Early Child Development
Keywords: Early Childhood Development; Unconditional Cash Transfer; Parenting; Randomized Controlled Trial; Women's empowerment; Household's decision making; Implementation science; Inequality

STUDY DESIGN:
Intervention Model Description: Clustered multi-arm Randomised Controlled Trial
Who Masked: Participant, Care Provider
Masking Description: Pregnant mothers and Community Health Workers will not know about the intervention arm they will be randomised to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (No Intervention): This group will serve as the Control group (81 HDs, 81 communities, 810 households) to identify the effects of a Parenting only, Unconditional Cash Transfer (UCT) only, and Parenting+UCT interventions. Caregivers will continue benefiting from a traditional government CHW home visit program, focusing on maternal and child health and nutrition, which is currently in practice in Tanzania.
- Parenting only (Experimental): 88 HDs, 77 communities, 770 households. Existing CHWs will be trained to use an innovative digital application for the delivery of integrated ECD services to mothers who are at least 20 weeks pregnant and less than 32 weeks pregnant for a period of 15 months. CHWs will provide tailored ECD services (e.g., prompting messages tailored to child age and triggering follow-up visits conditional on changing conditions), covering all aspects of the Nurturing Care Framework (Health, Nutrition, Responsive Caregiving, Early Learning, Safety and Security (WHO, UNICEF, World Bank Group, 2018)). Real time data will be recorded by the CHWs in each visit using the application. Data will include information on visit attendance, activities conducted, home environment, caregiver practices, and CHW observations. From when the target child is 6 months old, group sessions will be organised by CHWs, focusing on caregiver-child interaction and stimulation activities.
  Interventions: Other: Digital application supported CHW Parenting Intervention
- Parenting+Unconditional Cash Transfer (Experimental): 88 HDs, 77 communities, 770 households. In addition to the Parenting Intervention, pregnant women in the study sample will receive a bi-monthly unconditional mobile money transfer of 77,000 TZS (33 USD) from 5-7 months pregnancy over a period of 15 months (7 transfers in total).
  Interventions: Other: Digital application supported CHW Parenting Intervention; Other: Unconditional Cash Transfer Intervention
- Unconditional Cash Transfer only fixed amount (Experimental): 89 HDs, 80 communities, 800 households. Households, in addition to the CHWs delivering health and nutrition services as usual, will receive a fixed bi-monthly unconditional mobile money transfer each of 109,000 TZS (47USD) from 5-7 months pregnancy over a period of 15 months (7 transfers in total). The transfer will be randomly assigned between mothers and fathers/spouses within each community, where in half of the eligible households, mothers will receive the transfer and in the other half, fathers/spouses (or household head where the father/spouse is not available) will receive the transfer.
  Interventions: Other: Unconditional Cash Transfer only Intervention fixed amount
- Unconditional Cash Transfer only vary amount (Experimental): 89 HDs, 75 communities, 375 households. In addition to the previous four main treatment arms, there is another UCT only treatment study group where the level of the cash amount varies across communities. Communities, in addition to the CHWs delivering health and nutrition services as usual, in this group will be randomised to receive one of the bi-monthly unconditional mobile money transfer amounts: 32,000 TZS (14USD), 77,000 TZS (33USD), 109,000 TZS (47USD) from 5-7 months pregnancy over a period of 15 months (7 transfers in total). The transfers will be randomly assigned between mothers and fathers/spouses within each community, where in half of the eligible households, mothers will receive the transfer and in the other half, fathers/spouses (or household head where the father/spouse is not available) will receive the transfer.
  Interventions: Other: Unconditional Cash Transfer only Intervention vary amount

INTERVENTIONS:
Other: Digital application supported CHW Parenting Intervention — All pregnant women served by the trained CHW will be invited to participate in the Parenting program, from when the mother is at least 20 weeks pregnant and less than 32 weeks pregnant with the target child for a period of 15 months. CHWs will visit pregnant women at least 3 times during their pregnancy and at least 16 times following delivery. In addition to the individual home visits, the CHWs will organise bi-weekly in-community group sessions for children aged 6-12 months and their primary caregivers, focusing on caregiver-child interaction and stimulation activities.
  The immediate supervisors Health Care Workers (HCWs) of the CHWs will be trained to closely monitor CHWs activities and progress made. HCWs and CHWs will in turn be supervised and supported by district level Council Health Management Team (CHMT).
  Parenting services will be provided to all target children of these eligible caregivers, irrespective of their learning or physical abilities.
  Arms: Parenting only; Parenting+Unconditional Cash Transfer
Other: Unconditional Cash Transfer only Intervention fixed amount — The fixed cost for delivering the Parenting only Intervention was calculated to be 32,000 TZS. This cost is added to the average of maximum and minimum amount transferred on a bi-monthly basis to similar pregnant women under TASAF: 77,000 TZS. Therefore, in the 'Unconditional Cash Transfer fixed amount' treatment arm, the transfer will be 109,000 TZS (32,000 TZS + 77,000 TZS).
  Arms: Unconditional Cash Transfer only fixed amount
Other: Unconditional Cash Transfer Intervention — Families will receive from 5-7 months pregnancy over a period of 15 months a bi-monthly unconditional cash transfer, which equals the average of maximum and minimum amount transferred on a bi-monthly basis to similar pregnant women under Tanzania Social Action Fund (TASAF), i.e., Tanzania's National Cash Transfer program.
  Arms: Parenting+Unconditional Cash Transfer
Other: Unconditional Cash Transfer only Intervention vary amount — The rationale for the levels of the varying UCT amounts is to keep them comparable with i) the bi-monthly cost of the parenting program per family, ii) the bi-monthly cash transfers disbursed under TASAF, and iii) the sum of the bi-monthly cost of the parenting program and the bi-monthly cash transfer disbursed under TASAF. The fixed cost for delivering the Parenting Intervention was calculated to be 32,000 TZS. This cost is added to the average of maximum and minimum amount transferred on a bi-monthly basis to similar pregnant women under TASAF: 77,000 TZS. Therefore, in the 'Unconditional Cash Transfer only vary amount' group, each of the amounts vary individually (32,000 TZS; 77,000 TZS; 109,000 TZS).
  Arms: Unconditional Cash Transfer only vary amount

SUMMARY:
Digital solutions can significantly improve the delivery of Early Childhood Development (ECD) services in Low- and Middle-Income Countries (LMICs). Traditional home-visits and community group-based parenting approaches require intense levels of training, mentoring and supervision of Community Health Workers (CHWs) that is difficult to sustain when transitioning to scale. Context relevant digital tools can support CHWs in delivering high-quality, respectful, and standardised multi-sectoral household ECD services by tailoring services to pregnant women and engaging male caregivers. This could have significant impacts on child development, including stimulation, speech and language development, nutrition, and cognition. Moreover, cash delivered through digital modes of payment is faster, safer, easier to administer, is scalable and has potential to empower women, influence parental investment and affect household decision making. The study will conduct a clustered multi-arm Randomised Controlled Trial (cRCT) targeting pregnant mothers across all 7 districts (and all 8 district councils) in the Dodoma region in Tanzania. Following the study sample for 15 months from 5-7 months pregnancy. The study will test and compare the causal effects of (i) a digitally supported Parenting Intervention delivered by CHWs, which aims to improve caregivers' access to quality ECD services; (ii) a mobile unconditional cash transfer which aims to relax financial resource constraints; and (iii) a digitally supported Parenting Intervention when combined with a mobile unconditional cash transfer. Findings from the study are expected to have important policy implications for the design of scalable ECD interventions targeting pregnant mothers in Tanzania and other LMIC settings.

DETAILED DESCRIPTION:
The study will randomly sample 258 public Health Dispensaries (with at least one officially registered Community Health Worker (CHW) working at the facility) across all 7 districts (and all 8 district councils) in the Dodoma region, Tanzania, to participate in a clustered multi-arm Randomised Controlled Trial (cRCT). The 258 Health Dispensaries (HDs) will be randomised to a (i) Control group (81 HDs) where CHWs deliver Early Childhood Development (ECD) services as per existing government guidelines, (ii) Parenting group (88 HDs) where existing CHWs will be trained to use an innovative digital application for the delivery of integrated ECD services for a period of 15 months, from 5-7 months pregnancy onwards and, (iii) an Unconditional Cash Transfer (UCT) only group (89 HDs) where CHWs deliver ECD services as per existing government guidelines but where the study sample of families will receive a bi-monthly UCT fixed amount of 109,000 TZS (equivalent to 47USD) for 15 months (7 transfers in total). The randomisation will be stratified by district council and by whether there is more than one community in the HD catchment area.

Within each of the HD catchment areas in the Control group, one village (in rural areas) or one 'mtaa' (in urban areas) served by the HD and where at least one officially registered CHW is available to work will be randomly sampled. For the 88 Parenting HDs and the 89 UCT only HDs, all villages/mtaas (with at least one available officially registered CHW) will be included in their catchment area to become part of the study. In total, that will give 390 study villages/mtaas in the study sample.

Within each of the selected study villages/mtaas, one CHW will be selected whose catchment area will become the geographic area of interest, i.e., the study community. The study community can be the entire village, a hamlet (sub-village) or an mtaa, depending on the size of the CHW's catchment area. This gives a total of 82 Control communities, 155 Parenting communities, and 155 UCT communities in the study.

Within the Parenting and UCT only study groups, then second layer of randomisation will be done. In the Parenting group (154 communities across 88 HDs), communities will be randomly assigned, stratified by HD, to either one of the following two treatment arms: (i) Parenting only (77 communities) and (ii) Parenting+UCT (77 communities) where the Parenting Intervention will be delivered along with a bi-monthly unconditional mobile money transfer of 77,000 TZS (33 USD) from 5-7 months pregnancy over a period of 15 months (7 transfers in total). In the UCT only group (155 communities across 89 HDs), study communities will be randomly assigned, stratified by HDs, to either one of two treatment arms: (i) UCT only fixed amount (80 communities) where families will receive a fixed bi-monthly cash transfers each of 109,000 TZS (47 USD) over a period of 15 months (7 transfers in total) and (ii) UCT only vary amount where 77 communities will be randomly allocated to one of the following bi-monthly UCT amounts: 32,000 TZS (14 USD), 77,000 TZS (33 USD), 109,000 TZS (47 USD) over a period of 15 months (7 transfers in total). In each of these two study arms, further randomisation will be done whether the mobile money transfer is given to the father/spouse or the mother.

10 eligible women per community will de randomly sampled to participate in the study, except the bi-monthly UCT vary amount group, where only 5 eligible women per community will be randomly sampled.

Such a design allows to assess the relative cost-effectiveness of the Parenting and/or UCT only fixed amount interventions, and indeed provide insights into the value of adding a parenting component to a social protection program such as the Tanzania Social Action Fund (TASAF).

Additionally, the study will also explore CHW performance, quality of care delivered and other fidelity indicators to analyse impacts based on implementation effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18 years or above, who are living in the select study communities and who are at least 20 weeks pregnant and less than 32 weeks pregnant at the time of the baseline data collection survey visit to the study community region, Tanzania.

Exclusion Criteria:

* Households without pregnant women aged 18 years or above, who are living in the select study communities and who are at least 20 weeks pregnant and less than 32 weeks pregnant at the time of the baseline data collection survey visit to the study community region, Tanzania.
* If the pregnancy does not result in a live birth after enrolment, the respondent will be excluded from the study at the time of endline survey.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3585 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Children's cognitive, speech and language development | Endline survey (after 15 months)
  Direct assessment and parental report will be combined. For direct assessment, the Bayley-III (Bayley, 2006) suitably adapted for Tanzanian context will be used. Cognition, receptive and expressive language subtests will be selected. For parental report, selected items of the CREDI (McCoy et al, 2018) for cognition, receptive and expressive language subtests and a short version of the MacArthur-Bates Communicative Development Inventory (Jackson, 2012) that measures expressive language will be used, both already adapted for Tanzania. Raw scores will be standardized within the study sample for analysis. The measurement of outcomes will be aggregated using SEM to get latent factor(s) that summarizes effectively the information given by the individual items. Direct assessment and parental reports will be combined as well as the different child development domains if the fit of the model(s) are better than using the original raw scoring techniques were higher scores mean better outcomes.
Children's nutritional status | Endline survey (after 15 months)
  Weight and height will be measured at the time of the follow-up survey to obtain the height-for-age-z-scores and weight-for-height-age-z-scores, standard measures outlined by WHO. Mid Upper Arm Circumference (MUAC) will be also collected (WHO, 2006). Scores will be standardized within the study sample for analysis, so all measures are in the same metric. The measurement of nutritional outcomes will be aggregated using Structural Equation Modeling (SEM) to get latent factor(s) that summarizes effectively the information given by the individual outcomes. Different nutritional outcomes will be combined if the fit of the model(s) are better than using the individual z-scores.

SECONDARY OUTCOMES:
Children's socio-emotional development | Endline survey (after 15 months)
  Direct assessment and parental report will be combined. For the direct assessment, the Griffiths Developmental Scale III (Griffiths, 1970) personal-social-emotional subtest, suitably adapted for the context, will be used. For the parental report, selected items of the Caregiver Reported Early Development Instruments (CREDI) (McCoy, Marcus and Gunther, 2018) for the socio-emotional subtest which is already adapted for Tanzanian context and is free to use will be used. Raw scores will be standardized within the study sample for analysis. The measurement of outcomes will be aggregated using SEM to get latent factor(s) that summarizes effectively the information given by the individual items. Direct assessment and parental reports will be combined if the fit of the model(s) are better than using the original raw scoring techniques were higher scores mean better outcomes.
Child rearing practices | 15 months starting with baseline (October-December 2022) and finishing with endline survey (January-March 2024)
  The presence of toys and learning materials in the house will be assessed together with parental involvement with the child, the child's routines and organisation of the child's time inside and outside the family house. This will be assessed using the Family Care Indicators, developed by UNICEF (FCI) (Kariger, et al, 2012), selected subscales of the Home Observation for the Measurement of the Environment (HOME) (Bradley, 2014) and the Parental Style (PSQ) (Bornstein et al, 1996) for assessing social and didactic interactions. The measurement of outcomes will be aggregated using SEM to get latent factor(s) that summarises the information given by the individual items on time and monetary parental investments.

CONTACTS AND LOCATIONS:
Locations (1):
- Dodoma, Dodoma, Dodoma, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Anonymised Individual Participant Data will be shared 4 years after the endline survey of the study or after publishing journal paper(s).
Supporting Information: Study Protocol, SAP
Time Frame: 4 years after endline survey or after publishing journal paper(s).

REFERENCES:
- [Background] McCoy, D.C., Marcus W., and Günther F., "Measuring early childhood development at a global scale: Evidence from the Caregiver-Reported Early Development Instruments," Early Childhood Research Quarterly, 10 2018, 45, 58-68.
- [Background] Jackson-Maldonado D. MacArthur-Bates Communicative Development Inventories. The Encyclopedia of Applied Linguistics. 2012 Nov 5.
- [Background] World Health Organization. WHO child growth standards: length/height-for-age, weight-for-age, weight-for-length, weight-for-height and body mass index-for-age: methods and development. World Health Organization; 2006.
- [Background] Griffiths RB, Wheeler JC. Critical points in multicomponent systems. Physical Review A. 1970 Sep 1;2(3):1047.
- [Background] Kariger P, Frongillo EA, Engle P, Britto PM, Sywulka SM, Menon P. Indicators of family care for development for use in multicountry surveys. J Health Popul Nutr. 2012 Dec;30(4):472-86. doi: 10.3329/jhpn.v30i4.13417. PMID 23304914
- [Background] Bradley, R. H, "The HOME environment," in Marc H. Bornstein, ed., Handbook of Cultural Development Science, New York: Psychology Press, 2014, pp. 505-530.
- [Background] Bornstein, M. H., Tamis-LeMonda, C. S., Pascual, L., Haynes, O. M., Painter, K., Galperín, C., & Pêcheux, M.-G. Ideas about parenting in Argentina, France, and the United States. International Journal of Behavioral Development, 1996, 19, 347-367. https://doi.org/10.1177/016502549601900207
- [Background] Bayley, N., Bayley scales of infant and toddler development. PsychCorp., Pearson, 2006.
- [Background] World Health Organization, United Nations Children's Fund, World Bank Group. Nurturing care for early childhood development: a framework for helping children survive and thrive to transform health and human potential. Geneva: World Health Organization; 2018. Licence: CC BY-NC-SA 3.0 IGO. https://apps.who.int/iris/bitstream/handle/10665/272603/9789241514064-eng.pdf

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT05598970/Prot_SAP_001.pdf